CLINICAL TRIAL: NCT03509051
Title: Prospective Study on the Vaccine Response to Meningococcal B Vaccine After Allogeneic Stem Cell Transplantation
Acronym: MENINGREF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K180302J
Record Dates: First submitted 2018-04-13; First posted 2018-04-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Hematopoietic Stem Cell Transplant; Meningococcal Vaccine
Keywords: Allogeneic stem cell transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B vaccination (Experimental): One intramuscular injection of Bexsero (multicomponent B vaccine) from 6 months after transplant. A second similar dose will be given 2 months later.
  Interventions: Biological: B vaccination

INTERVENTIONS:
Biological: B vaccination — One intramuscular injection of Bexsero (multicomponent B vaccine) from 6 months after transplant. A second similar dose will be given 2 months later.

SUMMARY:
Allogeneic hematopoietic stem cell transplant (HSCT) recipients are at risk of various bacterial infections, especially due to a progressive decrease of specific antibodies. Around 90% of HSCT recipients have unprotective titers of specific antibodies to serogroups A and C meningogocci (Parkkali 2001; Mahler 2012).

Some small studies suggest that the response to meningococcal A and C vaccines is close to 100% after 3 doses given 18 months after transplant. Although the response to 2 doses of 4CMenB is over 75% in other immunocompromised patients (Feavers, 2017), studies with 4CMenB are lacking after HSCT. Nevertheless, as serogroup B caused 74% of IMD in Europe between 2004-2014 (Whittaker, 2017), the meningococcal B vaccination is recommended by the more recent guidelines from 6 months after transplant. There are, however, no data on the safety and efficacy of this vaccine after hematopoietic stem cell allograft (HSCT).

The objective of this study is to assess the response to 2 doses of a multicomponent meningococcal B vaccine (4CMenB) given at 2 months interval in adult allogeneic HSCT recipients transplanted at least 6 months ago.

The response will be assessed 1 month and 10 months after the second dose of vaccine by measuring bactericidal antibodies against NadA, fHbp, NHBA and PorAP1 vaccinal antigens according to methods previously reported (Caron Lancet Infect Dis 2011). The response rate will be correlated to pre- and post-transplant factors.

The hypothesis of this study is that 80% of the patients should have protective titers one month after the 2nd dose.

DETAILED DESCRIPTION:
Monocentric study. Forty patients are expected.

Primary objective: Response rate one month after 2 doses of vaccine

Secondary objectives: safety, rate of protection before vaccination, comparison of the antibody titers at one month vs. at 10 months after the vaccine program. Relationship between pre and post-transplant factors.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT at least 6 months before
* Age ≥ 18 years
* Platelet count > 50 G/L

Exclusion Criteria:

* Rituximab administration in the previous 6 months
* Relapse of the underlying disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
% of patients with Bactericidal titers > 4 to at least one component of the Bexsero vaccine, 1 month after the 2nd dose. | 1 month
  Vaccine response rate at one month after the 2nd dose.

SECONDARY OUTCOMES:
% of patients with Bactericidal titers > 4 to at least one component of the Bexsero vaccine, 12 months after the 1st dose. | 12 month
  Vaccine response rate at 12 month after the 1st dose.
Number of adverse events of vaccination by Bexsero after Allograft of CSH. | 12 month
  Number of adverse events (non serious and serious) reported during the study

CONTACTS AND LOCATIONS:
Overall Officials: Christine Robin, MD, Principal Investigator — Assistance Publique des Hopitaux de Paris
Locations (1):
- Henri-Mondor Hospital, Créteil, Val De Marne, France

REFERENCES:
- [Background] Caron F, du Chatelet IP, Leroy JP, Ruckly C, Blanchard M, Bohic N, Massy N, Morer I, Floret D, Delbos V, Hong E, Revillion M, Berthelot G, Lemee L, Deghmane AE, Benichou J, Levy-Bruhl D, Taha MK. From tailor-made to ready-to-wear meningococcal B vaccines: longitudinal study of a clonal meningococcal B outbreak. Lancet Infect Dis. 2011 Jun;11(6):455-63. doi: 10.1016/S1473-3099(11)70027-5. Epub 2011 Apr 12. PMID 21489881
- [Background] Mahler MB, Taur Y, Jean R, Kernan NA, Prockop SE, Small TN. Safety and immunogenicity of the tetravalent protein-conjugated meningococcal vaccine (MCV4) in recipients of related and unrelated allogeneic hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Jan;18(1):145-9. doi: 10.1016/j.bbmt.2011.07.027. Epub 2011 Aug 4. PMID 21820392
- [Background] Parkkali T, Kayhty H, Lehtonen H, Ruutu T, Volin L, Eskola J, Ruutu P. Tetravalent meningococcal polysaccharide vaccine is immunogenic in adult allogeneic BMT recipients. Bone Marrow Transplant. 2001 Jan;27(1):79-84. doi: 10.1038/sj.bmt.1702742. PMID 11244441
- [Background] Rubin LG, Levin MJ, Ljungman P, Davies EG, Avery R, Tomblyn M, Bousvaros A, Dhanireddy S, Sung L, Keyserling H, Kang I; Infectious Diseases Society of America. 2013 IDSA clinical practice guideline for vaccination of the immunocompromised host. Clin Infect Dis. 2014 Feb;58(3):309-18. doi: 10.1093/cid/cit816. PMID 24421306
- [Background] Whittaker R, Dias JG, Ramliden M, Kodmon C, Economopoulou A, Beer N, Pastore Celentano L; ECDC network members for invasive meningococcal disease. The epidemiology of invasive meningococcal disease in EU/EEA countries, 2004-2014. Vaccine. 2017 Apr 11;35(16):2034-2041. doi: 10.1016/j.vaccine.2017.03.007. Epub 2017 Mar 14. PMID 28314560